CLINICAL TRIAL: NCT03006692
Title: Diagnostic Value of Arterial Blood Gas Analysis in Prehospital Patients
Acronym: ABL
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stine Zwisler, Anesthesiologist, ph.d., Odense University Hospital
Other Study IDs: ABL Laegebil Odense
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Unconscious (Psychology)
MeSH Terms: conditions — Unconsciousness | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Take arterial blood gas: Patients with impaired consciousness are randomised into having analysed a arterial blood gas.
  Interventions: Other: With arterial blood gas, parameters not being normal can be corrected
- Do not take arterial blood gas: Patients with impaired consciousness are randomised into not having analysed a arterial blood gas.

INTERVENTIONS:
Other: With arterial blood gas, parameters not being normal can be corrected — If arterial blood gas is analysed answers provide the possibility to make more accurate diagnosis and treat specific abnormal parameters (e.g. electrolytes, oxygenation and so forth).
  Groups: Take arterial blood gas

SUMMARY:
In the anesthesiologist-manned mobile emergency car unit an analyzing device for blood gas testing is present since 2014. This study will determine if a prehospital arterial blood gas helps the doctor to make more precise diagnosis prehospitally. Furthermore it will be determined if the doctors find this device helpful in assessing and treating patients with affected consciousness.

ELIGIBILITY:
Inclusion Criteria:

* GCS < 13

Exclusion Criteria:

* Pregnant or breastfeeding
* detained or imprisoned patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 220 patients seen prehospital by the mobile emergency care unit in Odense, Denmark. Patients have to have impaired consciousness (Glasgow Coma Scale < 13).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 220 patients in 1.5 year
  Will there be fewer observational diagnosis

SECONDARY OUTCOMES:
Doctor satisfaction | 220 patients in 1.5 year
  Did the doctor find the arterial gas or lack of it affected the treatment and diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Odense, Denmark

REFERENCES:
- [Derived] Zwisler ST, Zincuk Y, Bering CB, Zincuk A, Nybo M, Mikkelsen S. Diagnostic value of prehospital arterial blood gas measurements - a randomised controlled trial. Scand J Trauma Resusc Emerg Med. 2019 Mar 18;27(1):32. doi: 10.1186/s13049-019-0612-8. PMID 30885262